CLINICAL TRIAL: NCT06610604
Title: Health-Related Quality of Life and Emotions in Patients with Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: Ming-an Yu (Other)
Responsible Party: Sponsor-Investigator, Ming-an Yu, Head of department of interventional medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: 17010406
Record Dates: First submitted 2024-09-02; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Nodule
Keywords: quality of life; anxiety; depression; spiritual health; thermal ablation; microwave ablation; thyroid nodules; papillary thyroid carcinoma
MeSH Terms: conditions — Thyroid Nodule; Anxiety Disorders; Depression; Thyroid Cancer, Papillary | interventions — Transurethral Resection of Prostate; Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- thyroidectomy: patients with thyroid nodules who undergo surgical resection
  Interventions: Procedure: thyroidectomy
- thermal ablation: patients with thyroid nodules who undergo thermal ablation
  Interventions: Procedure: thermal ablation

INTERVENTIONS:
Procedure: thermal ablation — thermal ablation including microwave ablation, radiofrequency ablation of thyroid nodules
  Groups: thermal ablation
Procedure: thyroidectomy — surgical resection of thyroid nodules
  Groups: thyroidectomy

SUMMARY:
The purpose of this observational research is to evaluate and compare the health-related quality of life and emotional well-being of patients with thyroid nodules before and after treatment. This is a data collection study by allowing investigators to access information generated before and after treatment.

DETAILED DESCRIPTION:
The incidence of thyroid nodules is rising worldwide. Papillary thyroid carcinoma (PTC), the most common type of thyroid cancer, has a favorable prognosis, with a low mortality rate and over 90% 10-year survival rate. Thyroidectomy is often applied to manage thyroid nodules as a traditional method. However, thermal ablation (TA), including microwave ablation (MWA), radiofrequency ablation (RFA), and laser ablation, has emerged as an alternative option for selected patients with thyroid function. TA methods are effective, safe, feasible, and have litter influence on thyroid function. Patients with thyroid nodules frequently exhibit higher levels of emotional stress compared to the general population. Additionally, health-related quality of life (QoL) has become an important endpoint and a strong predictor of survival time in medical and health research, underscoring the importance of treatments that not only prolong life but also preserve or enhance QoL. Considering the long survival time of patients with thyroid noduls and the similar therapeutic outcomes between surgery and MWA , it is crucial to pay more attention on patients' QoL and emotional well-being before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of benign thyroid nodules or papillary thyroid carcinoma ;
* underwent microwave ablation or thyroidectomy;
* ability to understand and cooperate with the survey

Exclusion Criteria:

* serious primary diseases in the liver, kidney, hematopoietic, or endocrine systems；
* a history of mental illness, personality disorders, cognitive impairments, or organic brain disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with thyroid nodules before and after treatments
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Thyroid Cancer-Specific Quality of Life Questionnaire to assess the thyroid-specific quality of life | before treatment and 1month, 6months, and 12 months after treatment
  The Thyroid Cancer-Specific Quality of Life Questionnaire (THYCA-QoL), as a methodologically developed questionnaire, was used to assess thyroid-specific symptoms in thyroid cancer survivors. The questionnaire consists of seven symptom scales (neuromuscular, voice, concentration, sympathetic, throat/mouth, psychological and sensory problems) and six single items (problems with scar, felt chilly, tingling hands/feet, gained weight, headache, less interest in sex), with a time frame of the previous week (except for less interest in sex item, which is four weeks), and each item is scored on a four-point response scale ranging from 1, "not at all", to 4, "very much". Scores were linearly transformed to a 0-100 scale. A higher score on this scale means more symptoms and complaints.
the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire to assess the general quality of life | before treatment and 1month, 6months, and 12 months after treatment
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) was adopted as a valid measurement of quality of life for cancer patients. It consists of 5 functional scales , 3 symptom scales, 6 single-item common symptom, and global health status (GHS) subscales. The time frame of the questions is the previous week, and each item is scored on a four-point response scale ranging from 1 to 4, except the global status scale, which is scored on a seven-point modified linear analog scale ranging from 1, "very poor" to 7, "excellent". After linear transformation, all scales and single item measures range in score from 0-100. A higher score on the functional scales and global status scale means a better level of functioning and HRQoL, whereas a a higher score on the symptom scales and single item corresponds to more discomfort and complaints.
Hospital Anxiety and Depression Scale to assess the emotional status | before treatment and 1month, 6months, and 12 months after treatment
  The Hospital Anxiety and Depression Scale consists of 14 items measuring symptom severity on a scale of 0-3 with subscales for anxiety (HADS_A) and depression (HADS_D), and a range of possible scores for each subscale of 0-21. Cut-off scores of 8+ for both subscales demonstrate the optimal balance between sensitivity and specificity for identifying cases of anxiety disorders and depression, with sensitivity and specificity of approximately .8 for both subscales.
The functional assessment of chronic illness therapy-spiritual well-being questionnaire to assess spiritual well-being | before treatment and 1month, 6months, and 12 months after treatment
  The functional assessment of chronic illness therapy-spiritual well-being scale consists of 12 items formatted in a five-point Likert scale ranging from 0 = not at all to 4 = very much, with the exception of two negatively stated items (4 and 8) coded in a reverse manner. The responses to the self-reported items refer to a 7-day recall period. The scores are added to generate a total score ranging from 0 to 48. With the highest scores representing better spiritual wellbeing.

SECONDARY OUTCOMES:
serum thyroid hormone | before treatment and 1month, 6months, and 12 months after treatment
  changes in serum thyroid hormone
Percent Volume Changes of Nodules | before treatment and 1month, 6months, and 12 months after treatment
  Percent Volume Changes of Nodules: ((Volume (baseline)- Volume (*m*))/Volume (baseline))*100

CONTACTS AND LOCATIONS:
Overall Officials: ming'an yu, MD, Study Chair — China-JapanFriendship Hospital
Locations (1):
- China-Japan Frienship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No